CLINICAL TRIAL: NCT05465798
Title: Beta-glucans as Immune Modulators Amongst Hospitalised Patients With COVID-19: A Pilot Randomised Trial
Brief Title: Beta-glucans for Hospitalised Patients With COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wohlstand Pharmaceutical (Industry)
Collaborators: Concentra Educación e Investigación Biomédica (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CON-001
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: beta-Glucans; Therapy; Signs and Symptoms; Mechanical ventilation; Inflammation; Survival
MeSH Terms: conditions — COVID-19; Signs and Symptoms; Inflammation

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomised to receive either beta-glucan supplements or placebo for up to three days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-Glucans (Experimental): Patients allocated to this arm will receive MC 3x3, an oral supplement containing 25mg of 1,3 beta-Glucans daily for up to three consecutive days.
  Interventions: Drug: MC 3x3
- Placebo (Placebo Comparator): Participants allocated to this arm will receive a placebo that will be identical in form to the MC 3x3 pills used the interventional arm. These doses will be scheduled daily and administered orally for up to three consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MC 3x3 — Patients allocated to this arm will receive MC 3x3, an oral supplement containing 25mg of 1,3 beta-Glucans of fungal origin (Trichoderma sp.) daily for up to three consecutive days.
  Arms: Beta-Glucans
Drug: Placebo — Patients allocated to this arm will receive a matching placebo similar to MC 3x3 pills used in the intervention arm. Placebos will be delivered orally every day for up to three consecutive days.
  Arms: Placebo

SUMMARY:
This randomised trial aims to assess the role of beta1-3 glucan supplementation in improving clinical symptoms and other outcomes amongst hospitalised patients with COVID-19.

DETAILED DESCRIPTION:
COVID-19 can present as a life-threatening disease characterised by respiratory failure and high circulating levels of inflammatory cytokines. Beta-glucans comprise a heterogeneous group of natural polysaccharides consisting of D-glucose monomers linked by a beta-glycosidic bond. They represent key structural elements of the cell wall and may serve as energy storage in bacteria, fungi including yeast, algae, and plants. In this triple-masked randomised trial, hospitalised patients requiring treatment with supplemental oxygen because of a laboratory-confirmed infection by SARS-CoV-2 will receive supplementation with 1-3 beta-glucans or placebo as part of their standard treatment. The primary endpoint of this trial is the intensity of clinical symptoms as detected by the Wisconsin Upper Respiratory Symptom Survey (WURSS).

Patients requiring mechanical ventilation at baseline will be excluded, as will those with cognitive impairment that precludes the use of clinical assessment scales, patients in which an order to limit therapeutic efforts has been issued, pregnant or breastfeeding women and those who decline to participate in this study. Secondary outcomes will include clinical deterioration requiring admission to an intensive care unit, requirement of high-flow nasal cannula or invasive mechanical ventilation and overall survival. Patients will be followed-up until hospital discharge or up to fifteen days after randomisation. Statistical analyses will be undertaken by a statistician unaware of treatment allocation under the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with an infection caused by SARS-CoV-2 confirmed with a reverse-transcription polymerase chain reaction (RT-PCR) obtained from a nasopharyngeal swab.

Exclusion Criteria:

* Life expectancy < 6 months
* Currently receiving invasive mechanical ventilation at baseline.
* Cognitive impairment that precludes the use of WURSS or understanding the informed consent form.
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Symptom severity | WURSS-21 scores calculated 1 day after randomisation
  Symptom severity based on the Wisconsin Upper Respiratory Symptom Survey (WURSS) score.
Symptom severity | WURSS-21 scores calculated 2 days after randomisation
  Symptom severity based on the Wisconsin Upper Respiratory Symptom Survey (WURSS) score.
Symptom severity | WURSS-21 scores calculated 3 days after randomisation
  Symptom severity based on the Wisconsin Upper Respiratory Symptom Survey (WURSS) score.
Symptom severity | WURSS-21 scores calculated 5 days after randomisation
  Symptom severity based on the Wisconsin Upper Respiratory Symptom Survey (WURSS) score.
Symptom severity | WURSS-21 scores calculated 7 days after randomisation
  Symptom severity based on the Wisconsin Upper Respiratory Symptom Survey (WURSS) score.
Symptom duration | Up to 2 weeks after randomisation or hospital discharge
  Total time with disease manifestations attributable to COVID-19.
Clinical recovery | Seven days after randomisation or up to hospital discharge
  Number of patients without clinical complaints attributable to COVID-19

SECONDARY OUTCOMES:
C-Reactive protein levels | This laboratory exam will be measured on days 1, 3, 5 and 7 after randomisation.
  C-Reactive protein levels measured at various time intervals during the hospitalisation.
Absolute lymphocyte count | This laboratory exam will be measured on days 1, 3, 5 and 7 after randomisation.
  Absolute lymphocyte counts measured at various time intervals during the hospitalisation.
Neutrophil to lymphocyte ratio | This laboratory exam will be measured on days 1, 3, 5 and 7 after randomisation.
  Neutrophil to lymphocyte ratios measured at various time intervals during the hospitalisation.
Intensive Care Unit Admission | Up to seven days after randomisation
  Proportion of patients requiring admission to an intensive care unit in each study group
Invasive mechanical ventilation | Up to seven days after randomisation
  Proportion of patients requiring invasive mechanical ventilation in each study group
Survival | Up to seven days after randomisation
  Proportion of patients that survived COVID-19 in each study group
Hospital Stay | Until hospital discharge
  Total stay within the hospital amongst participants

OTHER OUTCOMES:
Adverse events | Up to seven days after randomisation
  Adverse events attributable to Beta-Glucan supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Correa, MD, Study Director — Hospital Geriátrico Paz de La Tarde; Maria José Ruz, Principal Investigator — Hospital Gustavo Fricke; Mario Reyes, Principal Investigator — Science & Cash Group SpA; Felipe Martinez, MD, MSc, Principal Investigator — Concentra Investigacion; Michael Araya, Principal Investigator — Hospital Gustavo Fricke
Locations (1):
- Hospital Gustavo Fricke, Viña del Mar, Región de Valparaíso, Chile

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Yuki K, Fujiogi M, Koutsogiannaki S. COVID-19 pathophysiology: A review. Clin Immunol. 2020 Jun;215:108427. doi: 10.1016/j.clim.2020.108427. Epub 2020 Apr 20. PMID 32325252
- [Background] Qin C, Zhou L, Hu Z, Zhang S, Yang S, Tao Y, Xie C, Ma K, Shang K, Wang W, Tian DS. Dysregulation of Immune Response in Patients With Coronavirus 2019 (COVID-19) in Wuhan, China. Clin Infect Dis. 2020 Jul 28;71(15):762-768. doi: 10.1093/cid/ciaa248. PMID 32161940
- [Background] De Marco Castro E, Calder PC, Roche HM. beta-1,3/1,6-Glucans and Immunity: State of the Art and Future Directions. Mol Nutr Food Res. 2021 Jan;65(1):e1901071. doi: 10.1002/mnfr.201901071. Epub 2020 Apr 27. PMID 32223047
- [Background] Zimmerman JW, Lindermuth J, Fish PA, Palace GP, Stevenson TT, DeMong DE. A novel carbohydrate-glycosphingolipid interaction between a beta-(1-3)-glucan immunomodulator, PGG-glucan, and lactosylceramide of human leukocytes. J Biol Chem. 1998 Aug 21;273(34):22014-20. doi: 10.1074/jbc.273.34.22014. PMID 9705343
- [Background] Li B, Allendorf DJ, Hansen R, Marroquin J, Ding C, Cramer DE, Yan J. Yeast beta-glucan amplifies phagocyte killing of iC3b-opsonized tumor cells via complement receptor 3-Syk-phosphatidylinositol 3-kinase pathway. J Immunol. 2006 Aug 1;177(3):1661-9. doi: 10.4049/jimmunol.177.3.1661. PMID 16849475
- [Background] Mah E, Kaden VN, Kelley KM, Liska DJ. Beverage Containing Dispersible Yeast beta-Glucan Decreases Cold/Flu Symptomatic Days After Intense Exercise: A Randomized Controlled Trial. J Diet Suppl. 2020;17(2):200-210. doi: 10.1080/19390211.2018.1495676. Epub 2018 Oct 31. PMID 30380356
- [Background] Talbott S, Talbott J. Effect of BETA 1, 3/1, 6 GLUCAN on Upper Respiratory Tract Infection Symptoms and Mood State in Marathon Athletes. J Sports Sci Med. 2009 Dec 1;8(4):509-15. eCollection 2009. PMID 24149590